CLINICAL TRIAL: NCT03981666
Title: Systematic Self-screening of Insomnia and Proposition of a Video-Based Cognitive Behavioral Therapy for Insomnia in Adults Cancer Patients and Survivors: A Pilot Study
Brief Title: Video-Based Cognitive Behavioral Therapy for Insomnia in Adults Cancer Patients and Survivors
Acronym: SLEEP-4-ALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A00260-55; 2017/2659 (Other: CSET number)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with insomnia (Experimental): adult outpatients with a localized or metastatic breast, colorectal, pulmonary or urological cancer
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — To patients who have given their consent for the self-screening, the research assistant will propose 3 questionnaires, which will be completed in the waiting room and returned the same day:
  * Ad hoc questionnaire for demographics and medical data;
  * Insomnia Severity Index (ISI, 7 items, Savard et al., 2005);
  * Edmonton Symptom Assessment System (ESAS, 10 items, Visual Analogue Scale, Bruera et al. 1991) assessing comorbidities as pain, dyspnea, anxiety or depression...
  The ISI scoring will be realized by the research assistant (in the research office) immediately after its completion.

SUMMARY:
SLEEP-4-ALL-1 is a pilot and ecological study corresponding to the developpement phase of a randomized controlled multicentric trial SLEEP-4-ALL-2. The main objective of this second study will be the validation of a stepped-care model in the treatment of persistant insomnia in cancer patients.

The primary objective of SLEEP-4-ALL-1 is to determine the acceptability of a self-screening for insomnia in cancer outpatients at Gustave Roussy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults outpatients at Gustave Roussy,
2. with a breast, colorectal, pulmonary or urological,
3. localized or metastatic cancer,
4. during or after their treatment,
5. able to readily read and understand French,
6. able to use informatic tools confidently and with Internet access at home,
7. who have signed a written informed consent form prior to any study specific procedures,
8. affiliated to a social security system or beneficiary of the same.

Exclusion Criteria:

1. Age > 85 years old,
2. patient receiving a cancer diagnostic during a consultation of announcement
3. with a WHO index of 3 or 4
4. severe cognitive impairements or psychiatric disorders which are incompatible with the conditions and the conduct of the study (understanding of the objectives, completion of the questionnaires)
5. simultaneous participation in another study of the same type
6. patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2019-02-10 (Actual)

PRIMARY OUTCOMES:
Acceptance rate of self-screening for insomnia | Up to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided